CLINICAL TRIAL: NCT05940636
Title: A Novel Combined Neuromodulation Therapy to Enhance Balance and Neuroplasticity After Incomplete SCI
Brief Title: A Novel Combined Neuromodulation Therapy to Enhance Balance and Neuroplasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kei Masani, Senior Scientist, Associate professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-5262
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries; Muscle Pareses; Fall
MeSH Terms: conditions — Spinal Cord Injuries; Paresis

STUDY DESIGN:
Intervention Model Description: Single-center, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES+TSCS (combined) neuromodulation group (Experimental): For the combined neuromodulation with VFT group, the sub-motor threshold, open-loop TSCS will be coupled with closed-loop FES of ankle muscles during VFT. For this purpose, 2 electrical stimulators, one for each leg will stimulate SOL and TA muscles bilaterally while open-loop tonic lumbar TSCS will be applied at an intensity producing paresthesia in most of the lower-limb dermatomes
  Interventions: Other: Activity-based rehabilitation+electrical stimulation
- FES group (Active Comparator): For the FES with VFT group, participants will receive visual feedback regarding their center of pressure location during four games with varying levels of difficulty and FES will be applied bilaterally to SOL and TA via a closed-loop system.
  Interventions: Other: Activity-based rehabilitation+electrical stimulation

INTERVENTIONS:
Other: Activity-based rehabilitation+electrical stimulation — Balance training will occur three times per week for four weeks, totaling 12 two-hour sessions. In both groups, you will be asked to stand on a force plate while playing visual feedback training (VFT) games as part of the standing balance training. A force plate is similar to a bathroom scale that you can stand on which measures your body sway during movement. Visual feedback training (VFT) is a type of activity that includes weight-shifting movements in the upright stance. VFT will be done in both groups. There will be different games as shown in figure 1 and the order of the games will be randomly chosen in each session. During each game, there will be targets that will be presented on the screen and you will have to navigate toward them . You will be able to rest between games as needed.

SUMMARY:
Many people with partial damages in their spinal cord (iSCI) have physical impairments such as muscle paralysis in legs which make standing balance difficult. Poor balance control often leads to falls, injuries, and hospitalization. Therefore, improvement of standing balance is an important therapeutic goal for these individuals. Our team has shown that a therapy called visual feedback training (VFT) can improve standing balance by allowing individuals with iSCI to actively participate and follow visual feedback of their body sway on a screen like a computer game. We have also found that the application of low-energy electrical pulses to weak muscles called functional electrical stimulation (FES) during VFT can enhance the training effects. Recently, transcutaneous spinal cord stimulation (TSCS) has been discussed as a promising technique to further promote the rehabilitation effects after SCI by enhancing the connectivity between the brain and spinal cord and within the spinal pathways. However, to date, the potential of combining the two techniques (TSCS+FES) to improve the standing balance remains unknown. In this study, through the completion of a clinical trial, we will investigate the effects of an intervention that combines lumbar TSCS with FES of ankle muscles during VFT on the functional and neurophysiological outcomes in individuals living with iSCI. Participants will be randomly allocated to receive combined TSCS with FES or FES alone during VFT for 12 training sessions over 4 weeks. We expect that the new therapy would further improve balance and strengthen the neural connections between the brain and muscles. The expected changes in the neural connections will be measured by recording electrical signals from the lower limb muscles following stimulation of the motor region of the brain. Results of this study will be used for a larger-scale study in people with iSCI to improve balance and reduce falls during their daily life activities.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled trial to test the effects of a novel neuromodulation program on balance performance and neuroplasticity in individuals with iSCI. Participants will be randomly assigned to 2 equal groups labeled as (1) FES with VFT, and (2) combined neuromodulation with VFT. They will complete 8 training sessions over 4 weeks (2 sessions/week). For the FES with VFT group, participants will receive visual feedback regarding their center of pressure location during four games with varying levels of difficulty and FES will be applied bilaterally to SOL and TA via a closed-loop system. Each exercise will be completed 3 times per training session. For the combined neuromodulation with VFT group, the sub-motor threshold, open-loop TSCS will be coupled with closed-loop FES of ankle muscles during VFT. For this purpose, 2 electrical stimulators, one for each leg will stimulate SOL and TA muscles bilaterally while open-loop tonic lumbar TSCS will be applied at an intensity producing paresthesia in most of the lower-limb dermatomes. The range of FES stimulation intensity will vary between the minimal contraction threshold and 80% of the maximal tolerable threshold for each participant during games depending on the instant location of the participant's center of pressure and the location of the desired target during the game. All dependent variables will be assessed prior, immediately after, and 6-weeks after the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A traumatic or non-traumatic, non-progressive motor iSCI [American Spinal Injury Association Impairment Scale (AIS) rating of C or D];
2. More than 1-year post-injury;
3. ≥18 years old;
4. BBS score <46;
5. Free of any other condition besides SCI that significantly affects walking or balance (e.g., no vestibular disorder, significant vision loss, stroke)

Exclusion Criteria:

1. Neurological lesion levels below T12 ;
2. Severe spasticity in the legs;
3. Contractures in the lower extremities that prevent achieving a neutral hip and ankle position, or extended knee;
4. Peripheral nerve damage in the legs (i.e. leg muscles unresponsive to electrical stimulation);
5. A pressure sore (>grade 2) on the pelvis or trunk where the safety harness is applied;
6. Pregnancy;
7. History of epilepsy;
8. Contraindications for electrical stimulation (i.e. implanted electronic device, active cancer or radiation in past months, epilepsy, skin rash/wound at a potential electrode site)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Mini-Balance Evaluation Systems Test (mini-BESTest) | pre- immidiately post- 6 weeks follow up
  evaluates different components of postural control including anticipatory, reactive postural control, sensory orientation, and dynamic gait. It has high test-retest reliability, concurrent and convergent validity in individuals with iSCI.
10-meter Walk Test (10MWT) | pre- immidiately post- 6 weeks follow up
  performance-based measure to assess mobility and walking speed over a short distance.
Motor evoked potentials (MEP) | pre- immidiately post- 6 weeks follow up
  To measure neuroplasticity, we will record changes in the MEPs for the SOL and TA induced by TMS over the leg representation of the motor cortex

SECONDARY OUTCOMES:
Activities-specific Balance Confidence (ABC) Scale | pre- immidiately post- 6 weeks follow up
  self-reported questionnaire that evaluates balance confidence while performing 16 different mobility tasks such as walking around the house, sweeping the floor, climbing up and down the stairs, walking on a ramp and negotiating escalators
Falls Efficacy Scale - International (FES-I) | pre- immidiately post- 6 weeks follow up
  16-item self-reported questionnaire that measures fear of falling during basic and demanding daily life activities

CONTACTS AND LOCATIONS:
Overall Officials: Kei Masani, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute-Lyndhurst Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No